CLINICAL TRIAL: NCT00798291
Title: Evaluation of AN777 in Elderly Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Abbott Nutrition
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK32
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2010-03-22 (Estimated); Status verified 2010-03

CONDITIONS: Aged
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ad lib diet/placebo (Placebo Comparator): Ad lib diet and control product placebo
  Interventions: Other: Ad lib diet and Control placebo
- Ad lib diet/AN 777 (Experimental): Ad lib diet and AN 777
  Interventions: Other: Ad lib diet and An 777
- Ad lib diet/placebo/exercise (Active Comparator): Diet ad lib; exercise; and placebo
  Interventions: Other: Ad lib diet/ placebo/ exercise
- Ad lib diet/ AN 777/ exercise (Experimental): Diet ad lib; AN 777; exercise
  Interventions: Other: Ad lib diet; AN 777; exercise

INTERVENTIONS:
Other: Ad lib diet and Control placebo — one packet with water two times a day
  Arms: Ad lib diet/placebo
Other: Ad lib diet and An 777 — one packet with water two times a day
  Arms: Ad lib diet/AN 777
Other: Ad lib diet/ placebo/ exercise — one packet with water two times a day; resistance training three times a week
  Arms: Ad lib diet/placebo/exercise
Other: Ad lib diet; AN 777; exercise — one packet with water two times a day; resistance training three times a week
  Arms: Ad lib diet/ AN 777/ exercise

SUMMARY:
To evaluate whether AN777 with or without exercise affects muscle mass change in elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (male or female) is at least 65 years of age
2. Subject has a Geriatric Nutritional Risk Index (GNRI)of 92 or over
3. Subject has Body Mass Index (BMI) > 20.0 but <30.0
4. Subject is ambulatory
5. Subject agrees to maintain current activity level

Exclusion Criteria:

1. Subject has undergone major surgery, less than 4 weeks prior to enrollment in the study
2. Subject has current active malignant disease, except basal or squamous cell skin carcinoma or carcinoma in situ of the uterine cervix
3. Subject has stated immunodeficiency disorder
4. Subject has stated history of diabetes
5. Subject has stated presence of partial or full artificial limb
6. Subject has stated kidney disease
7. Subject has stated history of uncontrollable hypertension
8. Subject had myocardial infarction within the last 3 months
9. Subject had recent antibiotic use (within 1 week prior to screening).
10. Subject has a history of allergy to any of the ingredients in the study products
11. Subject has an obstruction of the gastrointestinal tract precluding ingestion of the study product, inflammatory bowel disease, short bowel syndrome or other major gastrointestinal disease
12. Subject has stated uncontrolled severe diarrhea, nausea or vomiting
13. Subject has untreated clinically significant ascites, pleural effusion or edema
14. Subject has known dementia, brain metastases, eating disorders, history of significant neurological or psychiatric disorder or any other psychological condition that may interfere with study product consumption
15. Subject is actively pursuing weight loss
16. Subject is currently taking medications/dietary supplements/substances that could profoundly modulate metabolism or weight Exceptions for multi-vitamin/mineral supplement, inhaled steroids for asthma or chronic obstructive pulmonary disease, topical or optical steroids and short-term use (less than two weeks) of dexamethasone

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the effect of AN777 on muscle mass change in an elderly population while on an adequate protein intake. | 24 weeks

SECONDARY OUTCOMES:
The secondary objective is to measure the effects of AN777 on body composition, functional outcomes, strength, and quality of life. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Johnson, PhD, Study Chair — Abbott Nutrition
Locations (1):
- Department of Health and Exercise Science, University of Oklahoma, Norman, Oklahoma, United States

REFERENCES:
- [Derived] Fukuda DH, Stout JR, Moon JR, Smith-Ryan AE, Kendall KL, Hoffman JR. Effects of resistance training on classic and specific bioelectrical impedance vector analysis in elderly women. Exp Gerontol. 2016 Feb;74:9-12. doi: 10.1016/j.exger.2015.12.002. Epub 2015 Dec 2. PMID 26657810
- [Derived] Stout JR, Fukuda DH, Kendall KL, Smith-Ryan AE, Moon JR, Hoffman JR. beta-Hydroxy-beta-methylbutyrate (HMB) supplementation and resistance exercise significantly reduce abdominal adiposity in healthy elderly men. Exp Gerontol. 2015 Apr;64:33-4. doi: 10.1016/j.exger.2015.02.012. Epub 2015 Feb 17. PMID 25700845